CLINICAL TRIAL: NCT00718302
Title: Ankle Fracture Plating: A Multicenter Randomized Trial Comparing Lateral and Antiglide Plating in Displaced Lateral Malleolus Fractures
Brief Title: A Multicenter Randomized Trial Comparing Antiglide and Lateral Plate Fixation in Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Paul Tornetta, III, M.D., Principal Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-27190
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Ankle Injuries
Keywords: Ankle Fractures; Displaced Lateral Malleolus Fractures; Antiglide Plating; Lateral Plating
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomized treatment; antiglide plate (Experimental): Randomized treatment; antiglide plate
  Interventions: Device: Antiglide Plate
- Randomized treatment; lateral plate (Experimental): Randomized treatment; lateral plate
  Interventions: Device: Lateral Plate

INTERVENTIONS:
Device: Antiglide Plate — A plate is placed behind the broken ankle and secured with screws
  Arms: Randomized treatment; antiglide plate
Device: Lateral Plate — A metal plate is placed to the side of the broken ankle and is secured with screws
  Arms: Randomized treatment; lateral plate

SUMMARY:
The role of operative fixation of unstable, displaced lateral malleolus fractures is well-established (Mayer, Mak, and Yablon). However, the optimal type of fixation remains the subject of debate. Lag screw fixation alone is only appropriate for long oblique fractures in younger patients (Tornetta). For all other patients, the choices for fibular stabilization most commonly involve the use of plates and screws which can be placed on either the lateral or posterior side of the bone, with or without lag screws. Lateral plating remains the most popular option, but since the description of posterior plating in 1982 (Brunner), reports in the literature have demonstrated some advantages of posterior over lateral plating (Ostrum, Treadwell, Winkler, and Wissing) . These advantages include less dissection, less palpable hardware, and decreased likelihood of intra-articular screw placement. However, there is only a single retrospective study in the published literature directly comparing these two methods (Lamontagne).

DETAILED DESCRIPTION:
Since it was first described in 1982, posterior antiglide plating has been presented as an attractive alternative to lateral plating of distal fibula fractures. Biomechanical studies have shown it to be a stronger construct than lateral plating, and other purported advantages include less dissection, decreased potential for intra-articular screw placement, and less palpable hardware decreasing the need for hardware removal.However, although posterior plating has become an accepted technique for operative management of these injuries, there is little clinical information in the literature regarding this treatment, and only one published retrospective study directly comparing posterior to lateral plating.

In 1996, Ostrum published a prospective study evaluating posterior plating in 32 patients, but only compared his results to a cohort of patients treated with lateral plating that was not part of his actual study group.Patel et al. recently presented a retrospective comparison of both techniques, but their study only included 29 patients in the lateral plating group and 23 in the posterior group.In both these studies, posterior plating was felt to be superior to lateral plating based on both the decrease in complications/re-operations related to symptomatic hardware, and improved function and pain scores.

However, in a much larger study, Lamontagneet al. showed no differences in operative time, complications or hardware removal rates in 193 patients reviewed retrospectively, and concluded that they could not recommend one treatment method over the other. They even elected not to proceed with a planned prospective study based on their results.A recent retrospective analysis of 70 patients showed a 43% incidence of need for hardware removal due to pain, with 30% of these patients having peroneal tendon lesions identified intra-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 85
* Closed Unstable Supination Eversion type Weber B fibula fracture
* Soft tissue amenable to operative treatment
* Opt for surgical treatment of their fracture
* Willing to follow up for 1 year
* Consent to be randomized

Exclusion Criteria:

* Aged < 18 or over 85
* Open fracture
* Prisoners
* Unlikely to followup
* Non english speaking
* Pre-existing arthrosis of the ankle
* Limitation in lower extremity function that would affect outcome scoring
* Significant anterior comminution precluding antiglide fixation
* Bilateral Fracture

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tornetta, MD, Principal Investigator — Boston University / Boston Medical Center; Laura Phieffer, MD, Principal Investigator — Ohio State University
Locations (10):
- United States (9):
  - Indiana University, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - New York Hospital for Joint Diseases, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma/ Health Science, Oklahoma City, Oklahoma
  - Orthopaedic Specialty Associates Fort Worth, Fort Worth, Texas
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 249 subjects were enrolled, but due to patient withdrawal or incomplete data from sites, only 233 subjects entered the flow.
Period: Overall Study
Arm/Group | Antiglide Plate | Lateral Plate
Started | 119 | 114
Completed | 119 | 114
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antiglide Plate | Lateral Plate | Total
Number analyzed (Participants) | 119 | 114 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 106 | 213
  >=65 years | 12 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Nonpalpable Hardware
Description: Percentage of Participants with Nonpalpable Hardware
Time Frame: 3 months, 6 months, 12 months
Population: Participants analyzed at 3 months - 88 (AP) / 89 (LP) Participants analyzed at 6 months - 68 (AP) / 67 (LP) Participants analyzed at 12 months - 53 (AP) / 51 (LP)
Measure: Number; unit: percentage of participants
Arm/Group | Antiglide Plate | Lateral Plate
Number analyzed (Participants) | 88 | 89
percentage of participants
  3 months | 71 | 55
  6 months: number analyzed (Participants) | 68 | 67
  6 months | 64 | 66
  12 months: number analyzed (Participants) | 53 | 51
  12 months | 51 | 44

2. Secondary Outcome: Percentage Normal Peroneal Tendons
Description: Percentage of Participants with Normal Peroneal Tendons
Time Frame: 3 months, 6 months, 12 months
Population: Participants analyzed at 3 months - 88 (AP) / 89 (LP) Participants analyzed at 6 months - 68 (AP) / 67 (LP) Participants analyzed at 12 months - 53 (AP) / 51 (LP) Numbers differ due to incomplete data collection or subjects were lost to follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Antiglide Plate | Lateral Plate
Number analyzed (Participants) | 88 | 89
percentage of participants
  3 months | 88 | 88
  6 months: number analyzed (Participants) | 68 | 67
  6 months | 91 | 92
  12 months: number analyzed (Participants) | 53 | 51
  12 months | 88 | 90

3. Secondary Outcome: American Orthopedic Foot and Ankle Society Score (AOFAS) Scores
Description: American Orthopedic Foot and Ankle Society Score (AOFAS) score. The questionnaire consists of nine items that are distributed over three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. A subject can score anywhere from 0-100, 100 being best.
Time Frame: 3 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antiglide Plate | Lateral Plate
Number analyzed (Participants) | 88 | 89
units on a scale
  3 months | 81.6 (12.8) | 82.8 (11.69)
  6 months: number analyzed (Participants) | 68 | 67
  6 months | 87.24 (10.74) | 87.43 (12.06)
  12 months: number analyzed (Participants) | 53 | 51
  12 months | 90.11 (9.52) | 89.44 (11.08)

4. Secondary Outcome: The Short Musculoskeletal Functional Assessment (SMFA) Score
Description: The Short Musculoskeletal Functional Assessment (SMFA) score. The questionnaire consists of four categories: Daily Activities, Emotional Status, Arm and Hand Function, Mobility. All categories are scored together, totaling between 0-100. The lower the score, the better the subjects function.
Time Frame: 3 months, 6 months, 9 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antiglide Plate | Lateral Plate
Number analyzed (Participants) | 88 | 89
units on a scale
  3 months | 25.1 (16.41) | 27.2 (19.36)
  6 months: number analyzed (Participants) | 68 | 67
  6 months | 15.3 (13.72) | 18.6 (18.75)
  12 months: number analyzed (Participants) | 53 | 51
  12 months | 11.6 (14.15) | 15.6 (17.6)

5. Secondary Outcome: SMFA - Bother Index
Description: The Bother Index is part of the SMFA. This section focuses on how much the injury is bothering the subject in terms of daily activities and use of injured area. The index totals are between 0-100. The lower the score, the less bothered the subject is by their injury.
Time Frame: 3 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Treatment; Antiglide Plate | Randomized Treatment; Lateral Plate
Number analyzed (Participants) | 88 | 89
units on a scale
  3 months | 23.1 (19.05) | 25.9 (20.07)
  6 months: number analyzed (Participants) | 68 | 67
  6 months | 14.1 (17.48) | 19.1 (20.09)
  12 months: number analyzed (Participants) | 53 | 51
  12 months | 12.8 (18.09) | 16.6 (22.04)

ADVERSE EVENTS:
Time Frame: 2 weeks, 6 weeks, 12 weeks, 26 weeks, 52 weeks
Arm/Group | Antiglide Plate | Lateral Plate
Serious Adverse Events (participants affected / at risk) | 1/119 | 1/114
Other Adverse Events (participants affected / at risk) | 13/119 | 8/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antiglide Plate (N=119) | Lateral Plate (N=114)
Non-Union (Surgical and medical procedures) | 0 (0) | 1 (1)
SUBJECT EXPIRED DUE TO CANCER (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antiglide Plate (N=119) | Lateral Plate (N=114)
PAINFUL IMPLANT-SCREW,PLATE (Surgical and medical procedures) | 4 (4) | 2 (2)
Infection (Infections and infestations) | 7 (7) | 2 (2)
Necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
DVT (Vascular disorders) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Developed Equinous Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loosening Hardware (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No